CLINICAL TRIAL: NCT01345968
Title: Preoperative Intravenous Ferric Carboxymaltose (Ferinject) in Patients With Orthopedic Surgery and High Risk of Blood Loss
Brief Title: Intravenous Ferric Carboxymaltose (Ferinject) in Patients Undergoing Orthopaedic Surgery
Acronym: PRIVIRON
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Less patients than expected for inclusion, therefore recruitment is too low
Sponsor: University Hospital Muenster (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UKM10_0027; 2010-024115-14 (EudraCT Number); 05-AnIt-09 (Other: Department of Anesthesiology and Intensive Care, University Hospital Muenster)
Record Dates: First submitted 2011-04-21; First posted 2011-05-02 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-07

CONDITIONS: Anemia; Orthopedic Surgery; High Risk of Blood Loss
Keywords: anemia; transfusion; intravenous ferric carboxymaltose
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NaCl 0.9% (Placebo Comparator)
  Interventions: Drug: NaCl 0.9%
- Ferinject (Experimental)
  Interventions: Drug: Ferinject 50 mg/ml

INTERVENTIONS:
Drug: Ferinject 50 mg/ml — iv administration of max. 50 ml (Dilution: 20 ml in 30 ml NaCl 0.9%) in 30 minutes
  Arms: Ferinject
Drug: NaCl 0.9% — iv administration of max. 50 ml in 30 minutes
  Arms: NaCl 0.9%

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of preoperative intravenous ferric carboxymaltose in patients with anemia undergoing hip or knee replacement

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* Patients scheduled to undergo hip or knee replacement
* 8 g/dl < Hb < 13 g/dl for men and 8 g/dl < Hb < 12 g/dl for women at screening (3-4 weeks prior to surgery)
* anemia
* signed written informed consent

Exclusion Criteria:

* immunosuppressive or myelosuppressive therapy
* history of thromboembolic events
* a concurrent medical condition(s) that would prevent compliance or participation or jeopardize the health of the patient
* hypersensitivity to any component of the formulation
* transfusion within 1 month prior to study inclusion
* liver values 3 times higher than normal
* active severe infection/inflammation
* renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Number of RBC units | Until postoperative day 7

SECONDARY OUTCOMES:
Blood transfusion rate | Until postoperative day 7
  Number of patients with blood transfusions
Frequency of postoperative complications | Until postoperative day 7
  Number of postoperative complications from baseline until postoperative day 7
Frequency of postoperative complications | Until 6 weeks after surgical intervention
  Number of postoperative complication from baseline until 6 weeks after surgical intervention
Length of hospital stay | 6 weeks after surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hugo K Van Aken, PhD, MD, Principal Investigator — Department of Anesthesia and Intensiv Care, University Hospital Muenster
Locations (2):
- Germany (2):
  - Charité Universitätsmedizin Berlin, Berlin
  - University Hospital Muenster, Münster